CLINICAL TRIAL: NCT06677827
Title: Effect of Adding Magnesium Sulphate As Adjuvant to Bupivacaine in Ultrasound Guided External Oblique Intercostal Plane Block in Upper Abdominal Cancer Surgery
Brief Title: Effect of Adding Magnesium Sulphate As Adjuvant to Bupivacaine in Ultrasound Guided External Oblique Intercostal Plane Block in Upper Abdominal Cancer Surgery.to Assess the Total Postoperative Opioid Consumption in the First 24 H and Evaluate Post Operative VAS Score
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Raghda Ramadan Ahmed, resident doctor at Anesthesia, Intensive Care and Pain Management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MgSO4 EOIB Abd Cancer Surgery
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Upper Abdominal Cancer Surgery
Keywords: External Oblique Intercostal Plane Block; Magnesium Sulphate; Bupivacaine
MeSH Terms: interventions — Bupivacaine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups Group 1: 20 ml bupivacaine 0.25%+200 mg magnesium sulphate Ultrasound guided external oblique intercostal plane block bilateral Group 2: 20 ml bupivacaine 0.25% only Ultrasound guided external oblique intercostal plane block bilateral
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent anesthesiologist randomly using computer-generated random numbers divided the patients into 2 groups :(Group 1 and Group 2). Each group will include 34 patients. We discreetly placed the randomization results in envelopes until the end of the study. The researchers who were responsible for postoperative follow-up and data processing were blinded to the group allocation during the whole study period. All patients were also blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group bupivacaine (Experimental)
  Interventions: Drug: Bupivacaine
- group magnesium sulphate &bupivacaine (Experimental)
  Interventions: Drug: Magnesium Sulfate and Bupivacaine 0.125%

INTERVENTIONS:
Drug: Bupivacaine — External Oblique Intercostal plane block technique with 20 ml bupivacaine 0.25% only bilateral
  Arms: group bupivacaine
Drug: Magnesium Sulfate and Bupivacaine 0.125% — External Oblique Intercostal plane block technique with 20 ml bupivacaine 0.25%+200 mg magnesium sulphate bilateral
  Arms: group magnesium sulphate &bupivacaine

SUMMARY:
double blind randomized controlled trial will be conducted on upper abdominal cancer surgery cases to study the effect of Adding Magnesium Sulphate as Adjuvant to Bupivacaine in Ultrasound Guided External Oblique Intercostal Plane Block in Upper Abdominal Cancer Surgery

DETAILED DESCRIPTION:
Despite advances in the field of medical and radiation oncology, surgical resection is a crucial intervention and remains the mainstay of gold standard treatment. Upper abdominal incisions such as the oblique subcostal laparotomy are a cause of severe pain and can lead to significant respiratory impairment . Numerous studies have demonstrated that when enhanced recovery procedures (ERPs) are used, hospital length of stay, time to return to normal function, postoperative ileus duration, thromboembolic complications, morbidity, and all of these factors are all reduced. Traditionally, epidural analgesia has been the cornerstone of pain control in such surgeries. However, it has limitations, including potential complications and contraindications in certain patients.

The innervation of the upper abdominal wall originates from the T6th and T10th intercostal nerves and requires effective blocking of these nerves to achieve analgesic and anesthetic efficacy. For upper abdominal surgeries, the ideal regional anesthesia technique should target both the anterior and lateral cutaneous branches of the intercostal nerves from T6 to T10. Hesham Elsharkawy et al demonstrated the potential mechanism of the external oblique intercostal fascial plane block (EOIB) in a cadaver study in which both lateral and anterior branches of the intercostal nerves T7-T10 were stained. Patients to whom this block was applied exhibited consistent dermatomal sensory blockade between T6-T10 in the anterior axillary line and T6-T9 in the midline. It has been shown that this block can be used in the clinical setting for upper abdominal wall analgesia. The external oblique intercostal (EOI) block has shown promising results in covering the anterior and lateral upper abdominal wall. It's simple, effective, and convenient block, particularly in the context of morbid obesity.

The external oblique intercostal block offers effective pain relief for the upper abdomen without the systemic effects of sympathetic blockade and without impairing motor or bladder function. It ensure optimal pain management, promote early postoperative mobilization, and support functional recovery.

Magnesium is a calcium blocker and an NMDA receptor antagonist. Research has demonstrated that magnesium sulfate [MgSO4] has an analgesic effect by blocking N-methyl-D-aspartate [NMDA] receptors and associated calcium channels, thereby preventing central sensitization that arises due to peripheral nociceptive stimulation. Magnesium may influence the central nervous system's (CNS) ability to transmit nociceptive signals and pain sensation in the central nervous system (CNS) by inhibiting N-methyl-D-aspartate (NMDA) receptor and calcium channels. It was used recently as a powerful analgesic adjuvant resulting in reduced postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* a. Age >18 years old b. Both sex c. Patients who were in risk-scoring groups I-III of the American Society of Anesthesiologists (ASA)

Exclusion Criteria:

* c. Patients' refusal, d. History of allergy to any of the study medications e. Any contraindications to regional anesthesia. f. Patients with anatomical abnormalities. g. Patients have hemodynamic instability. h. Patients with local infection, and suspected intra-abdominal sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
dose postoperative opioid consumption | baseline
  the total dose postoperative opioid consumption in the first 24 h.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] El Sherif F, Gomaa Sayed D, Fares KM, Mohamed SA, Osman AM, Kamal Sayed A, Mamdouh Kamal S. Magnesium Sulfate in Pediatric Abdominal Cancer Surgery: Safety and Efficacy in Ultrasound-Guided Transversus Abdominis Plane (US-TAP) Block in Conjugation with Levobupivacaine. Local Reg Anesth. 2023 Sep 12;16:133-141. doi: 10.2147/LRA.S425649. eCollection 2023. PMID 37719936
- [Background] Cosarcan SK, Ercelen O. The analgesic contribution of external oblique intercostal block: Case reports of 3 different surgeries and 3 spectacular effects. Medicine (Baltimore). 2022 Sep 9;101(36):e30435. doi: 10.1097/MD.0000000000030435. PMID 36086688
- [Background] Mehmet Selim C, Halide S, Erkan Cem C, Onur K, Sedat H, Senem U. Efficacy of Unilateral External Oblique Intercostal Fascial Plane Block Versus Subcostal TAP Block in Laparoscopic Cholecystectomy: Randomized, Prospective Study. Surg Innov. 2024 Aug;31(4):381-388. doi: 10.1177/15533506241256529. Epub 2024 May 23. PMID 38780355
- [Background] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112
- [Background] Korkusuz M, Basaran B, Et T, Bilge A, Yarimoglu R, Yildirim H. Bilateral external oblique intercostal plane block (EOIPB) in patients undergoing laparoscopic cholecystectomy: A randomized controlled trial. Saudi Med J. 2023 Oct;44(10):1037-1046. doi: 10.15537/smj.2023.44.10.20230350. PMID 37777270
- [Background] Lin T, Yu J, Hu Y, Liu H, Lu Y, Zhao M, Chen H, Chen X, Li G. [Preliminary experience of dual-port laparoscopic distal gastrectomy for gastric cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2019 Jan 25;22(1):35-42. Chinese. PMID 30703792